CLINICAL TRIAL: NCT02365805
Title: Randomized Open-label, Multicentric, Phase II Clinical Trial to Evaluate the Efficacy of a Neoadjuvant Chemotherapy Scheme Customized by Levels of BRCA1 in Women With Primary HER2 Negative Breast Cancer (The BERNAQ Clinical Trial)
Brief Title: Randomized CT to Evaluate Efficacy of Neoadjuvant Chemotherapy Customized by Levels of BRCA1-HER2 Negative Breast Cancer
Acronym: BERNAQ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-005843-28
Record Dates: First submitted 2014-12-30; First posted 2015-02-19 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
Keywords: BRCA 1 levels; HER2 Negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Cyclophosphamide; Fluorouracil; Paclitaxel; Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard FEC Regimen (Active Comparator): Epirubicin + Ciclofosfamide + Fluorouracil + Paclitaxel
  Interventions: Drug: Epirubicin + Ciclofosfamide + Fluorouracil + Paclitaxel
- No or Low BRCA1 expression (Experimental): Epirubicin + Cisplatin + Fluorouracil
  Interventions: Drug: Epirubicin + Cisplatin + Fluorouracil
- Normal or High BRCA1 expression (Experimental): Docetaxel + Ciclofosfamide
  Interventions: Drug: Docetaxel + Ciclofosfamide

INTERVENTIONS:
Drug: Epirubicin + Ciclofosfamide + Fluorouracil + Paclitaxel — Epirubicin 90 mg/m2 + Ciclofosfamide 600 mg/m2 + 5-Fluorouracil 600 mg/m2 intravenous infusion on day 1 every three weeks, for four cycles; followed by Paclitaxel 100 mg/m2 weekly for eight weeks.
  Other Names: Standard FEC Regimen
  Arms: Standard FEC Regimen
Drug: Epirubicin + Cisplatin + Fluorouracil — Epirubicin 60 mg/m2 + Cisplatin 60 mg/m2 intravenous infusion on day 1 every three weeks and 5-Fluorouracil 200 mg/m2/day for eight cycles.
  Other Names: QT combination
  Arms: No or Low BRCA1 expression
Drug: Docetaxel + Ciclofosfamide — Docetaxel 75 mg/m2 + Ciclofosfamide 600 mg/m2, intravenous infusion on day 1 every three weeks, for eight cycles.
  Other Names: QT combination
  Arms: Normal or High BRCA1 expression

SUMMARY:
Neoadjuvant chemotherapy (NAC) is increasingly used for early-stage operable breast cancer. Response of breast cancer to NAC is correlated with survival: patients who obtain greatest survival advantage are those who attain complete response of their primary tumor. BReast Cancer 1 (BRCA1) plays a crucial role in DNA repair and associations between BRCA1 mRNA expression and sensitivity to platinum and/or resistance to taxanes has been previously documented. We propose a two-arm, randomized, multi-centre, open-label phase II study to compare the efficacy and tolerability of NAC customized by BRCA 1 levels versus standard FEC chemotherapy, being pathological complete response the primary endpoint.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy (NAC) is increasingly used for early-stage operable breast cancer. Response of breast cancer to NAC is correlated with survival: patients who obtain greatest survival advantage are those who attain complete response of their primary tumor.BReast Cancer 1 (BRCA1) plays a crucial role in DNA repair. Associations between BRCA1 mRNA expression and sensitivity to platinum and/or resistance to taxanes are previously documented. Improving complete response rates with NAC we can improve outcomes in breast cancer. If we establish biomarkers which predict better response we may optimized treatment by individualized breast cancer care. Therefore, we propose a two-arm, randomized, multi-centre, open-label phase II study. The study will compare the efficacy and tolerability of NAC customized by BRCA 1 levels versus standard chemotherapy, being pathological complete response the primary endpoint. Women with primary Her-2 negative breast cancer who have not undergone previous treatment for invasive breast cancer will be randomized to receive the following: Treatment Arm 1 (standard therapy): 5-Fluorouracil, Epirubicin and Cyclophosphamide day 1 every 3 weeks per three cycles; Treatment Arm 2: Patients with low levels of BRCA1 mRNA will receive Epirubicin and Cisplatin day 1 every 3 weeks and 5-Fluorouracil for three cycles; And patients with high levels of BRCA1 will receive docetaxel day 1 every three weeks per three cycles. Definitive surgery will be performed within 4 weeks after the last cycle.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* 18 years or older
* Performance Status- ECOG: 0-1
* Histologically confirmed invasive breast cancer
* Primary tumor greater than 2 cm diameter
* Any N (0-3)
* No evidence of metastasis (M0), HER-2/ERBb2 negative.
* Known hormone receptors status.
* Haematopoietic status: Absolute neutrophil count > 1.5 x 109/L; Platelet count > 100 x 109/L
* Hemoglobin at least 9 g/dl)
* Hepatic status: Serum total bilirubin < 1.5 x upper limit of normal (ULN), in the case of known Gilbert's syndrome, a higher serum total bilirubin (< 2 x ULN) is allowed;AST and ALT < 2.5 times ULN; Alkaline phosphatase < 2.5 times ULN)
* Renal status: Creatinine < 1.5 mg/dl or Cl CR > 60 ml/m
* For women of childbearing potential Negative serum pregnancy test, within 2-weeks (preferably 7 days) prior to randomization.
* Signed informed consent form (ICF).

Exclusion Criteria:

* Received any prior treatment for primary invasive breast cancer.
* Previous (less than 10 years) or current history of malignant neoplasms, except for curatively treated:
* Basal and squamous cell carcinoma of the skin;Carcinoma in situ of the cervix.
* Diagnosis of inflammatory breast cancer.
* Known history of uncontrolled or symptomatic angina, clinically significant arrhythmias, congestive heart failure, transmural myocardial infarction uncontrolled hypertension (? 180/110), unstable diabetes mellitus, dyspnoea at rest, or chronic therapy with oxygen.
* Left Ventricular Ejection Fraction of < 50% measured by echocardiography.
* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical disorder that would interfere with the subject?s safety.
* Unresolved or unstable, serious adverse events from prior administration of another investigational drug.
* Active or uncontrolled infection.
* Dementia, altered mental status, or any psychiatric condition that would prevent the understanding or rendering of ICF.
* Concurrent neoadjuvant cancer therapy (chemotherapy, radiation therapy, immunotherapy, biologic therapy other than the trial therapies).
* Concurrent treatment with an investigational agent or participation in another therapeutic clinical trial.
* Known immediate or delayed hypersensitivity reaction, idiosyncrasy or contraindication to drugs chemically related to any of the study treatments or their excipients.
* Pregnant or lactating women.
* Refusal to use contraception throughout the study (surgical sterilization, barrier methods associated with spermicidal gels or total abstinence). Use of hormonal contraceptives is not allowed.
* Patient unable to comply with study procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2016-10-10 (Actual); Study Completion 2016-10-10 (Actual)

PRIMARY OUTCOMES:
Rate of residual tumor types RCB-0 and RCB-I (good pathological response) at the time of surgery. | 4-8 weeks after the last neoadjuvant chemotherapy cycle.
  To evaluate and compare the rate of good pathological response (residual tumor types RCB-0 and RCB-I) at the time of surgery in patients with ER or PgR positive, or triple negative (non-Her2/Erb 2 overexpressing and/or amplified) breast cancer randomized to standard neoadjuvant chemotherapy (NAC) based in anthracyclines versus customized NAC according levels of BRCA1 expression.

SECONDARY OUTCOMES:
Percentaje of patients candidates to conventional mastectomy as indicated by surgeon | At baseline and after the last neoadjuvant chemotherapy cycle (up to 24 weeks after randomization).
Rates of residual tumor types RCB-0, RCB-I, RCB-II and RCB-III pathological response in surgical breast and axillary node resection specimens | 4-8 weeks after the last neoadjuvant chemotherapy cycle .
Percentage of patients with negative axillary nodes | 4-8 weeks after the last neoadjuvant chemotherapy cycle.
Complete tumoral response at the time of surgery (WHO criteria). | At baseline and after the last neoadjuvant chemotherapy cycle (up to 24 weeks after randomization).
Percentaje of patients candidates to breast conserving mastectomy as indicated by surgeon | At baseline and after the last neoadjuvant chemotherapy cycle (up to 24 weeks after randomization).
Partial tumoral response at the time of surgery (WHO criteria). | At baseline and after the last neoadjuvant chemotherapy cycle (up to 24 weeks after randomization).

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Ruiz-Borrego, MD, Principal Investigator — University Hospital Virgen del Rocío
Locations (7):
- Spain (7):
  - Hospital Universitario Puerta del Mar, Cadiz, Cádiz
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - Hospital Universitario Juan Ramón Jimenez, Huelva, Huelva
  - Complejo Hospitalario de Jaén, Jaén, Jaén
  - Hospital Universitario Virgen Macarena, Seville, Seville
  - Hospital Universitario Virgen del Rocío, Seville, Seville
  - Hospital Universitario Nuestra Señora de Valme, Seville, Seville